CLINICAL TRIAL: NCT06715137
Title: Microvascular Dysfunction in Adults with Congenital Heart Disease and the Effect of Exercise Training
Acronym: MICONEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Edge 001475
Record Dates: First submitted 2024-11-26; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Congenital Heart Defect; Congenital Heart Disease; Microvascular Dysfunction; Exercise Training; Oxidative Stress; Coronary Microvascular Dysfunction; Peripheral Microvascular Dysfunction
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Exercise; Resistance Training

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise arm (Experimental): Each participant received a personalized rehabilitation schedule combining aerobic interval cycle training and a dynamic strength exercise program, developed to ensure that the participants met the physical activity guidelines.
  Interventions: Behavioral: Exercise training
- Conventional care arm (No Intervention): In the conventional care arm, patients did not receive explicit exercise advice but were provided with general information regarding a healthy lifestyle, in accordance with current physical activity guidelines during the first study visit.

INTERVENTIONS:
Behavioral: Exercise training — Each participant received a personalized rehabilitation schedule combining aerobic interval cycle training and a dynamic strength exercise program, developed to ensure that the participants met the physical activity guidelines. For the aerobic training, the patients cycled for 30-45 minutes on an exercise bike at home 3 times a week. During each training session, the heart rate (HR) was continuously recorded using a chest strap and displayed in a smartphone application. The target HR zones were predefined with alternating intervals of intensive and extensive aerobic training. The program followed a progressive structure with the objective of completing 40 minutes of intensive aerobic training after 16 weeks. In the strength training program, 4 dynamic exercises targeting major muscle groups were performed 3 times a week. Every 2 weeks, these exercises were intensified by altering the starting position or adding extra weight.
  Other Names: Exercise program; Home-based aerobic and strength exercise program; Training program; Exercise training progam
  Arms: Exercise arm

SUMMARY:
The goal of this prospective cohort study is to deepen the understanding of the pathophysiology in adults with congenital heart disease (CHD). Through this research, the investigators aim to identify potential strategies to improve the prevention and treatment of these patients. In this context, the effects of exercise training will also be assessed. The main questions it aims to answer are:

* Is coronary microvascular dysfunction (MVD) present in adults with diverse types of CHD?
* Is peripheral MVD present in adults with diverse types of CHD?
* Are coronary and peripheral MVD correlated in adults with diverse types of CHD?
* Is microvascular function correlated with inflammation and oxidative stress in adults with diverse types of CHD?
* Are inflammation and oxidative stress correlated with ventricular function in adults with diverse types of CHD?
* Are MVD and diminished ventricular function interrelated and associated with reduced exercise capacity in adults with diverse types of CHD?
* Does exercise training in adults with CHD result in improvements in coronary and peripheral microvascular function, inflammation and oxidative stress, biventricular function, muscle strength, exercise capacity and quality of life?

For the last research question, patients were randomized to receive either conventional care or home-based aerobic and strength exercise training.

ELIGIBILITY:
Inclusion Criteria:

* adults with congenital heart disease: as many different types of CHD as possible were incorporated
* New York Heart Association (NYHA) class I-II
* who visited the out-patient clinic at the Antwerp University Hospital

Exclusion Criteria:

* smoking
* body mass index >35 kg/m²
* professional endurance athlete
* the presence of macrovascular coronary artery disease
* diabetes mellitus
* a systemic disease (e.g., malignancies, acute and chronic inflammatory diseases in the preceding 3 months)
* a contraindication for adenosine administration.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Coronary microvascular function: coronary flow reserve | on both study visits (at baseline and at 16 weeks)
  The coronary flow reserve (CFR) was measured using pulsed wave Doppler measurements at the mid to distal left anterior descending artery (LAD) in an apical modified 2-chamber view. At baseline and during hyperemia (following a 3-minute period of intravenous adenosine administration at a rate of 140 µg/kg/min), three optimal profiles of peak diastolic Doppler flow velocities were measured, and the results were averaged. CFR was then calculated as the ratio between hyperemic and basal average peak velocities.

SECONDARY OUTCOMES:
Peripheral microvascular function: reactive hyperemia index | on both study visits (at baseline and at 16 weeks)
  Peripheral microvascular function was measured by peripheral arterial tonometry (PAT)(Endo-PAT2000®, Itamar Medical, software version 3.2.4, Caesarea, Israel). Relative ischemia was provoked by inflating a blood pressure cuff on the forearm to a minimum of 100 mmHg above systolic blood pressure. Following a 5-minute period, reactive hyperemia was induced by rapidly deflating the cuff. The reactive hyperemia index (RHI) is defined as the ratio of the average amplitude of the PAT signal over a one-minute period starting one minute after cuff deflation (maximum pulse amplitude) divided by the average amplitude of the PAT signal over a 3.5 minute period preceding cuff inflation (baseline pulse amplitude). RHI and Framingham modified RHI (fRHI) were calculated by dedicated software (Itamar Medical).
Peripheral microvascular function: Framingham modified reactive hyperemia index | on both study visits (at baseline and at 16 weeks)
  Peripheral microvascular function was measured by peripheral arterial tonometry (PAT)(Endo-PAT2000®, Itamar Medical, software version 3.2.4, Caesarea, Israel). Relative ischemia was provoked by inflating a blood pressure cuff on the forearm to a minimum of 100 mmHg above systolic blood pressure. Following a 5-minute period, reactive hyperemia was induced by rapidly deflating the cuff. The reactive hyperemia index (RHI) is defined as the ratio of the average amplitude of the PAT signal over a one-minute period starting one minute after cuff deflation (maximum pulse amplitude) divided by the average amplitude of the PAT signal over a 3.5 minute period preceding cuff inflation (baseline pulse amplitude). RHI and Framingham modified RHI (fRHI) were calculated by dedicated software (Itamar Medical).
Carotid arterial wall thickness: carotid intima-media thickness | on both study visits (at baseline and at 16 weeks)
  The carotid intima-media thickness (IMT) was measured: B-mode and color Doppler ultrasound, equipped with a 10 MHz linear array transducer (Aloka Prosound 6 Ultrasound Linear Probe LN 5413, Hitachi Aloka Medical, Japan) was used to evaluate the right common, internal and external carotid arteries. A standardized protocol was applied to evaluate carotid IMT: briefly, all subjects were examined in a supine position with their head turned 45 degrees from the site being scanned. Measurements were made using automated e-tracking of the wall along a distance of 2 cm. Three measurements were taken at the common carotid artery, approximately 2 cm proximal to the carotid bifurcation, and the values were averaged to determine the mean IMT.
Large artery stiffness: pulse wave velocity | on both study visits (at baseline and at 16 weeks)
  Systemic large artery stiffness was measured using pulse wave velocity (PWV) and augmentation index (AIx)(Sphygmocor system®, AtCor Medical, West Ryde, Australia).
  For PWV, an applanation tonometer (Millar Instruments) was positioned on both the right common carotid artery and the right femoral artery. Proximal (i.e., carotid) and distal (i.e., femoral) pulses were recorded consecutively and were averaged. PWV was calculated as the carotid-to-distal path length divided by the transit time. In order to prevent overestimation, a scaling factor of 0.8 was applied to convert PWV values obtained using the direct carotid-femoral distance to the corrected PWV (PWVc).
Large artery stiffness: augmentation index | on both study visits (at baseline and at 16 weeks)
  Systemic large artery stiffness was measured using pulse wave velocity (PWV) and augmentation index (AIx)(Sphygmocor system®, AtCor Medical, West Ryde, Australia).
  For central AIx, three measurements were obtained using the applanation tonometer (Millar Instruments) at the level of the right carotid artery. AIx was determined as the ratio of augmentation (which is attributed to wave reflection) to pulse pressure (defined as the difference between systolic and diastolic pressure).
Inflammation: white blood cell count | on both study visits (at baseline and at 16 weeks)
  Fasting peripheral blood was collected using ethylenediaminetetraacetic acid (EDTA) tubes (BD Vacutainer®, Canada). EDTA samples were analyzed using a Sysmex XN-9100 (Sysmex, Germany) to quantify white blood cell counts.
Inflammation: high-sensitivity C-reactive protein | on both study visits (at baseline and at 16 weeks)
  Fasting peripheral blood was collected using serum vacuette tubes (BD Vacutainer®, Canada). Serum samples were analyzed using an Atellica® IM/CH Analyzer (Siemens Healthcare, Germany) to quantify high-sensitivity C-reactive protein (hs-CRP) concentrations.
Oxidative stress: superoxide anion radical | on both study visits (at baseline and at 16 weeks)
  Superoxide anion radical levels were quantified using electron paramagnetic resonance (EPR) spectroscopy.
  When fasting venous blood samples from the patients were obtained in a heparin tube (BD vacutainer®, Canada), 100 µl of blood was immediately added to 100 µL of spin probe CMH. Immediately after mixing, the sample was snap frozen and stored at -80°C until analysis. For analysis conducted at the University of Maastricht (Department of Toxicogenomics), the mixture of CMH and blood was thawed and transferred into a 50 μl glass capillary (Hirschmann®, Germany). The glass capillaries were placed in the resonator of the EPR. EPR measurements were carried out on a Bruker EMX 1273 spectrometer equipped with an ER 4119HS high-sensitivity resonator and 12 kW power supply operating at X band frequencies. The data were analyzed using WinEPR (Brüker, Germany) software and radicals were identified and quantified as ESR peak amplitude arbitrary units (A.U.).
Left ventricular function: ejection fraction | on both study visits (at baseline and at 16 weeks)
  All echocardiographic examinations were performed by two experienced sonographers utilizing harmonic imaging on an EPIQ7 ultrasound system (Philips Medical Systems, Best, the Netherlands). A detailed 2D transthoracic echocardiogram was performed with the patient placed in the left lateral decubitus position.
  For the assessment of left ventricular (LV)* systolic function, LV ejection fraction (LVEF) was measured using the Simpson biplane method.
  * The term "LV" refers to the morphological LV
Left ventricular function: global longitudinal strain | on both study visits (at baseline and at 16 weeks)
  All echocardiographic examinations were performed by two experienced sonographers utilizing harmonic imaging on an EPIQ7 ultrasound system (Philips Medical Systems, Best, the Netherlands). A detailed 2D transthoracic echocardiogram was performed with the patient placed in the left lateral decubitus position.
  For the assessment of left ventricular (LV)* systolic function, LV global longitudinal strain (LV GLS) was calculated by combining 3 apical longitudinal LV chamber views (2-, 3- and 4-chamber).
  * The term "LV" refers to the morphological LV
Right ventricular function: fractional area change | on both study visits (at baseline and at 16 weeks)
  The right ventricle (RV)* was comprehensively assessed using the novel two-dimensional multiplane echocardiography (2D MPE) approach revealing 4 RV views: a focused, non-foreshortened RV view (4C), coronary sinus view (CS), aortic view (Ao) and coronal view (CV).
  RV fractional area change (FAC)(calculated as: (end-diastolic-end-systolic area)/end-diastolic area x100) was recorded in all 4 RV views. In addition to the values from the individual RV walls, a multiwall average was computed when measurements from at least 3 walls of one individual were feasible to obtain.
  * The term "RV" refers to the morphological RV
Right ventricular function: tricuspid annular plane systolic excursion | on both study visits (at baseline and at 16 weeks)
  The right ventricle (RV)* was comprehensively assessed using the novel two-dimensional multiplane echocardiography (2D MPE) approach revealing 4 RV views: a focused, non-foreshortened RV view (4C), coronary sinus view (CS), aortic view (Ao) and coronal view (CV).
  RV tricuspid annular plane systolic excursion (TAPSE)(measured with 2D echocardiography-guided M-mode) was recorded in all 4 RV views. In addition to the values from the individual RV walls, a multiwall average was computed when measurements from at least 3 walls of one individual were feasible to obtain.
  * The term "RV" refers to the morphological RV
Right ventricular function: tissue Doppler imaging systolic velocity | on both study visits (at baseline and at 16 weeks)
  The right ventricle (RV)* was comprehensively assessed using the novel two-dimensional multiplane echocardiography (2D MPE) approach revealing 4 RV views: a focused, non-foreshortened RV view (4C), coronary sinus view (CS), aortic view (Ao) and coronal view (CV).
  RV tissue Doppler imaging systolic velocity (TDI S') was recorded in all 4 RV views. In addition to the values from the individual RV walls, a multiwall average was computed when measurements from at least 3 walls of one individual were feasible to obtain.
  * The term "RV" refers to the morphological RV
Right ventricular function: peak systolic global longitudinal strain | on both study visits (at baseline and at 16 weeks)
  The right ventricle (RV)* was comprehensively assessed using the novel two-dimensional multiplane echocardiography (2D MPE) approach revealing 4 RV views: a focused, non-foreshortened RV view (4C), coronary sinus view (CS), aortic view (Ao) and coronal view (CV).
  Peak systolic global longitudinal RV strain (RV LS) was assessed in 3 of the 4 RV views (i.e., 4C, CS, Ao) using an automated strain software (AutoStrain; Philips Medical Systems, Best, the Netherlands). In each RV view, a single RV free wall strain value was derived from the average of 3 segments (basal, mid and apical). A multiwall average was calculated if at least 2 RV free walls were feasible to measure.
  * The term "RV" refers to the morphological RV
Quality of life: RAND 36-Item Health Survey 1.0 | on both study visits (at baseline and at 16 weeks)
  The patients were asked to complete a quality of life questionnaire consisting of a combination of the RAND 36-Item Health Survey 1.0 and the EuroQol visual analogue scale (EQ-VAS).
  The RAND 36-Item Health Survey 1.0 encompasses 8 health domains: physical functioning, bodily pain, role limitations due to physical health issues, role limitations due to personal or emotional concerns, general mental health, social functioning, energy/fatigue, and general health perception. Additionally, it incorporates a single item aimed at assessing perceived change in health.
Quality of life: EuroQol visual analogue scale | on both study visits (at baseline and at 16 weeks)
  The patients were asked to complete a quality of life questionnaire consisting of a combination of the RAND 36-Item Health Survey 1.0 and the EuroQol visual analogue scale (EQ-VAS).
  The EQ-VAS is a vertical scale to self-rate the patients' current health state, ranging from 0 (worst imaginable) to 100 (best imaginable).
Exercise capacity: percent-predicted peak oxygen consumption | on both study visits (at baseline and at 16 weeks)
  A cardiopulmonary exercise test was conducted until maximal exhaustion. Therefore, a continuously incrementing ramp protocol (increase of work rate, e.g., every 2-15 seconds) was implemented with the objective of achieving maximal exertion within 8-12 minutes using a Lode Corival bike ergometer. The protocol was chosen based on the Jones' predictions of maximal power output. Throughout the test, gas exchange measurements and 12-lead electrocardiogram readings were continuously recorded, while blood pressure was monitored every minute. Peak oxygen consumption (pVO2) was determined as the mean VO2 during the final 30 seconds of exercise. Subsequently, percent-predicted peak oxygen consumption (%ppVO2) was computed, using the reference values following Wasserman et al. and the LowLands registry.
Muscle strength: one-repetition maximum | on both study visits (at baseline and at 16 weeks)
  The one-repetition maximum (1RM) was measured for 4 different exercises targeting major muscle groups: chest press, vertical traction, low row, and leg press (BioCircuit Series 4, TechnoGym®, Benelux).

CONTACTS AND LOCATIONS:
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vanreusel I, Vermeulen D, Goovaerts I, Stoop T, Ectors B, Cornelis J, Hens W, de Bliek E, Heuten H, Van Craenenbroeck EM, Van Berendoncks A, Segers VFM, Briede JJ. Circulating Reactive Oxygen Species in Adults with Congenital Heart Disease. Antioxidants (Basel). 2022 Nov 30;11(12):2369. doi: 10.3390/antiox11122369. PMID 36552576
- [Background] Vanreusel I, Taeymans J, Van Craenenbroeck E, Segers VFM, Van Berendoncks A, Briedé JJ, et al. Oxidative Stress in Patients with Congenital Heart Disease: A Systematic Review. Advances in Redox Research. 2024:100109
- [Background] Vanreusel I, Taeymans J, Van Craenenbroeck E, Segers VFM, Van Berendoncks A, Briede JJ, Hens W. Elevated oxidative stress in patients with congenital heart disease and the effect of cyanosis: a meta-analysis. Free Radic Res. 2023 May-Jun;57(6-12):470-486. doi: 10.1080/10715762.2023.2284639. Epub 2023 Dec 26. PMID 38000042
- [Background] Vanreusel I, Hens W, Van Craenenbroeck E, Van Berendoncks A, Segers VFM. Peripheral Microvascular Dysfunction in Children and Adults with Congenital Heart Disease: A Literature Review. Curr Cardiol Rev. 2024;20(4):e210224227260. doi: 10.2174/011573403X278440240209064408. PMID 38409710
- [Background] Vanreusel I, Segers VFM, Craenenbroeck EV, Berendoncks AV. Coronary Microvascular Dysfunction in Patients with Congenital Heart Disease. Curr Cardiol Rev. 2023;19(4):e190123212886. doi: 10.2174/1573403X19666230119112634. PMID 36658708